CLINICAL TRIAL: NCT04510688
Title: Study of the Effectiveness and Safety of Cabozantinib Treatment in Patients With Advanced Renal Cell Carcinoma (RCC) Under a Spanish Managed Access Program and Real-world Practice
Brief Title: Spanish Real-World Evidence Cabozantinib
Acronym: SRWEC
Status: Completed | Type: Observational
Sponsor: Spanish Oncology Genito-Urinary Group (Other)
Collaborators: Syntax for Science, S.L (Industry); Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: SOGUG-2017-A-IEC(REN)-7
Record Dates: First submitted 2020-06-29; First posted 2020-08-12 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — cabozantinib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Managed Access Program (MAP) patients: Patients with RCC treated with cabozantinib under a Managed Access Program (MAP) prior to Cabometyx® marketing authorization
  Interventions: Drug: Cabozantinib
- Real World (RW) patients: Patients with RCC treated with cabozantinib as routine clinical prescription (Real World), with treatment started after Cabometyx® marketing authorization
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — Observation of treatment with Cabozantinib

SUMMARY:
RCC (Renal Cell Carcinoma) is the most common form of kidney cancer, accounting for 2-3% of all adult malignancies and for 90% of all kidney cancers. The incidence of RCC has steadily increased over the past two decades, showing a plateau in recent years. Many patients with RCC remain asymptomatic until late disease stages and other patients have disease at diagnosis (metastatic RCC or mRCC).

Recently, the tyrosine kinase inhibitor (TKI) cabozantinib was approved as a first-line therapy for patients with advanced clear-cell RCC (ccRCC). Cabozantinib was initially approved for patients previously treated with antiangiogenic therapy based on the phase 3 METEOR study, which demonstrated a clinical benefit compared with everolimus.

Immunotherapy has been also developed in ccRCC.

The frontline treatment paradigm for ccRCC has evolved, particularly for intermediate-/poor-risk patients, with the recent addition of cabozantinib and nivolumab/ipilimumab (immunotherapy), but overall survival data are needed to understand their benefit-to-risk profiles compared with established therapies.

In October 2016, the Spanish Agency of medicines (AEMPS) granted the temporary Authorization for special use to Cabometyx® 20/40/60 mg within a Managed Access Program (MAP) for the treatment of advanced RCC in adults following prior VEGF-targeted therapy (Vascular Endothelial Growth Factor targeted therapy). The MAP allows the possibility of using a medicinal product which is not yet commercially available or approved. By the end of the MAP period, on July 2017, 136 patients had been included by 61 centers who received at least one dose of Cabometyx® for the treatment of advanced RCC.

Since then, Cabometyx® 20/40/60 mg was made commercially available for the treatment of advanced RCC in adults following prior VEGF-targeted therapy. After the commercialization of Cabometyx® in July 2017 in Spain, the inclusion of new patients in the MAP was closed but those patients that were already included continued receiving Cabometyx® free of charge until clinical decision. In July 2018, the European Commission approved a new indication for adult patients previously untreated with intermediate or poor risk.

Based on this rationale, the aim of this study is to obtain safety and effectiveness information regarding the use of cabozantinib in a non-selected RCC population, both in patients that received this agent under the MAP or under routine clinical prescription (real-world [RW]).

ELIGIBILITY:
Inclusion Criteria:

1. Male or females, aged 18 years or older.
2. Diagnosis of advanced Renal Cell Carcinoma (RCC)
3. Alive or dead patients at study initiation who received at least one dose of cabozantinib for the treatment of RCC between October 2016 and 1 st June 2019.
4. Alive patients who agree to participate and signed the Informed Consent Form (ICF).

Exclusion Criteria:

1. Patients who decline consent.
2. Patients whose hospital medical records are unavailable for review.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data from patients with Renal Cell Carcinoma (RCC) currently under tretament at the study site or data from deceased patients with RCC
Sampling Method: Non-Probability Sample
Enrollment: 275 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Effectiveness: Progression-Free Survival | Through study completion, an average of 2 years
  Evaluation of the effectiveness of cabozantinib in terms of investigator-assessed PFS (Progression-Free Survival) based on the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
Incidence of Adverse Reactions | Through study completion, an average of 2 years
  Evaluation of the safety of cabozantinib by recording the incidence of adverse reactions in both MAP and RW cohorts.
Incidence of dose reductions | Through study completion, an average of 2 years
  Evaluation of the safety of cabozantinib by recording the incidence of dose reductions in both MAP and RW cohorts.
Incidence of temporary interruptions or discontinuations | Through study completion, an average of 2 years
  Evaluation of the safety of cabozantinib by recording the Incidence of temporary interruptions or discontinuations in both MAP and RW cohorts.
Incidence of use of medications to manage adverse reactions | Through study completion, an average of 2 years
  Evaluation of the safety of cabozantinib by recording the incidence of use of medications to manage adverse reactions in both MAP and RW cohorts.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Suárez, MD, Principal Investigator — Investigator
Locations (32):
- Spain (32):
  - Hospital Universitario Reina Sofía, Córdoba, Andalusia
  - Hospital Universitario Juan Ramón Jiménez, Huelva, Andalusia
  - Complejo Hospitalario de Jaén, Jaén, Andalusia
  - Hospital Son Llatzer, Palma de Mallorca, Balearic Islands
  - Hospital Universitari Parc Taulí, Sabadell, Barcelona
  - Hospital Unviersitario de Gran Canaria Doctor Negrin, Las Palmas de Gran Canaria, Canary Islands
  - Hospital Universitario Nuestra Señora de Candelaria, Santa Cruz de Tenerife, Canary Islands
  - Hospital Universitario de León, León, Castille and León
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Hospital Universitari Sant Joan de Reus, Reus, Catalonia
  - Consorci Corporació Sanitària Parc Taulí de Sabadell, Sabadell, Catalonia
  - Hospital Universitario de Badajoz, Badajoz, Extremadura
  - Centro Oncológico de Galicia, A Coruña, Galicia
  - Complejo Hospitalario Universitario de Ferrol, Ferrol, Galicia
  - Complejo Hospitalario Universitario Ourense, Ourense, Galicia
  - Hospital Universitari Son Espases, Palma de Mallorca, Illes Ballears
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Clínico Universitario de Valenica, Valencia, Valencia
  - Hospital Universitari Dr. Peset, Valencia, Valencia
  - Hospital Universitari i Politècnic La Fe, Valencia, Valencia
  - Hospital Del Mar, Barcelona
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital Provincial de Castellón, Castellon
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital General de Ciudad Real, Ciudad Real
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Virgen de La Salud, Toledo
  - Fundación Instituto Valenciano de Oncología, Valencia
  - Hospital Arnau de Vilanova, Valencia
  - Hospital Universitario Alvaro Cunqueiro, Vigo

IPD SHARING:
Plan to Share IPD: No